CLINICAL TRIAL: NCT07051954
Title: Investigation of the Effects of Functional Respiratory Muscle Training on Respiratory Muscle Function, Exercise Capacity, Skeletal Muscle Strength, and Muscle Endurance in Individuals With Post-COVID-19 Syndrome
Brief Title: Effectiveness of Functional Respiratory Muscle Training in Post-COVID-19 Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/12-16
Record Dates: First submitted 2025-07-03; First posted 2025-07-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Post COVID-19 Syndrome; Functional Inspiratory Muscle Training; Core Stabilization
Keywords: Post-COVID Syndrome; Trunk Muscle Endurance; Exercise Capacity; Functional Inspiratory Muscle Training (IMT); Core Stabilization
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: The study includes two groups: one group performing core stabilization exercises and the other performing both core stabilization and functional inspiratory muscle training.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization Group (Active Comparator): Participants will receive an 12-week core stabilization exercise program only.
  Interventions: Other: Core Stabilization
- Functional IMT Group (Experimental): Participants will receive an 12-weeks core stabilization exercise program plus functional inspiratory muscle training (IMT).
  Interventions: Other: Core Stabilization; Other: Functional Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Other: Core Stabilization — 12-week supervised core stabilization training, 3 sessions per week, 45 minutes per session.
Other: Functional Inspiratory Muscle Training (IMT) — IMT using a portable inspiratory muscle training device at 60% MIP, progressively increased over 12 weeks.
  Arms: Functional IMT Group

SUMMARY:
This study aims to investigate the effects of core stabilization exercises and functional inspiratory muscle training (IMT) on various physiological and psychological parameters in individuals with post-COVID-19 syndrome. Participants diagnosed with post-COVID-19 syndrome will be randomly assigned to two groups using stratified computer-assisted randomization. One group will undergo an 8-week core stabilization training, while the other will receive combined core stabilization and IMT training. Exercise training will be conducted three times a week, with each session lasting 50 minutes.

Comprehensive pre- and post-intervention assessments will be conducted, including exercise capacity, respiratory and peripheral muscle strength, trunk endurance, balance, anxiety, depression, and fatigue levels. The primary outcome measures are respiratory muscle strength and trunk endurance.

Participants must be aged 18-65 years, have at least a primary education level, speak Turkish, and be classified as level 2-3 on the Post-COVID-19 Functional Status Scale (PCFS). Eligible participants will be referred by the Internal Medicine Department at Hacettepe University.

The study will utilize various assessment tools, including maximal inspiratory/expiratory pressure (MIP/MEP) tests, Functional Movement Screen (FMS), plank and Sorenson endurance tests, the Timed Up and Go Test for balance, handgrip and knee extension strength tests, body composition analysis, and the SF-36 quality of life questionnaire.

DETAILED DESCRIPTION:
This study aims to investigate the effects of core stabilization programs supported by core stabilization exercises and functional inspiratory muscle training (IMT) on various physiological and psychological parameters in individuals with post-COVID-19 syndrome.

Participants to be included in the study will consist of individuals diagnosed with post-COVID syndrome and will be divided into two groups with a computer-aided stratified randomization method.

After the patients are randomly separated, one group will receive 8 weeks of core stabilization training and the other group will receive functional IMT (IMT combined with core stabilization) training. The exercise program is designed to last 8 weeks in total, and the training program for both groups will be carried out on certain days (3 days) per week, and each session will last 50 minutes.

A comprehensive assessment will be applied to both groups at the beginning and end of the study. These assessments are; exercise capacity, respiratory muscle strength, peripheral muscle strength, trunk muscle endurance, balance, anxiety and depression levels, and fatigue level parameters. The primary outcome measure of the study will be respiratory muscle strength and trunk muscle endurance.

Individuals who meet the inclusion criteria will be included in the study. The study will be conducted with individuals between the ages of 18-65, with at least primary school education, and whose local language is Turkish. Participants diagnosed with Post-COVID-19 Syndrome and who are in class 2-3 according to the Post-COVID-19 Functional Status Scale (PCFS) will be included in the study. Participants who are eligible for the study will be directed to the Cardiopulmonary Rehabilitation Unit of the Hacettepe University Faculty of Physical Therapy and Rehabilitation by the relevant physicians of the Department of General Internal Medicine of the Hacettepe University Department of Internal Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Post-COVID-19 Syndrome.
* Literate and able to understand study procedures.
* Aged between 18 and 65 years.
* Willing to voluntarily participate in the study.
* Classified as functional class 2-3 according to the Post-COVID-19 Functional Status Scale (PCFS).
* Clinically stable; comorbid conditions such as hypertension or diabetes must be controlled.
* No orthopedic or neurological conditions that would prevent assessment of peripheral muscle strength, balance, or exercise capacity.

Exclusion Criteria:

* History of recent myocardial infarction or pulmonary embolism.
* Presence of uncontrolled chronic diseases.
* Any orthopedic or neurological disorders that limit mobility.
* Neurological impairments (e.g., cerebrovascular disease) or psychiatric disorders that impair cooperation or compliance with exercise testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | Baseline and after 12 weeks of intervention.
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) with mouth-pressure device
Plank Endurance Test | Baseline and after 12 weeks of intervention.
  Plank Test: Plank time is a common test to evaluate core stability. The patient is given a plank position and the maximum endurance time they can hold this position is measured.
Sorenson Endurance Test | Baseline and after 12 weeks of intervention.
  Sorenson Test (Extensor Endurance Test): In this test, the person lies horizontally on the end of a table and is asked to keep their body in a fixed position outside the table. The endurance time in this position is evaluated to measure core stability.
Side Bridge Endurance Test | Baseline and after 12 weeks of intervention.
  Side Bridge Test: It is an endurance test based on time in the side plank position. The difference between the times on the right and left sides can provide information about core stabilization.

SECONDARY OUTCOMES:
Health Status | Baseline and after 12 weeks of intervention.
  The Short-Form-36 is a quality of life questionnaire consisting of 11 sections and 36 questions in total. The minimum and maximum scores range between 0 and 100. Higher score indicate a more favorable health status.
Fatigue Perception | Baseline and after 12 weeks of intervention.
  Fatigue Severity Scale consists of 9 questions that indicate severity of fatigue in daily life. The total score 4 and more indicate the presence of severe fatigue and ranges between 0-7.
Dynamic respiratory muscle strength | Baseline and after 12 weeks of intervention.
  In the dynamic method, respiratory muscle strength index (S index) and peak inspiratory flow rate (PIF) will be assessed using the portable POWERbreathe K5 device (PowerBreathe K5, HaB International Ltd, Warwickshire, England).
Exercise motivation | Baseline and after 12 weeks of intervention.
  Patients' exercise motivation levels and attitudes will be assessed with the Exercise Motivation Attitude Questionnaire. The Exercise Motivation Attitude Scale consists of 20 items and three subscales. The total score that can be obtained from the scale ranges from 20 to 140 (minimum 20, maximum 140). The score varies depending on the number of items in the subscales. Higher scores indicate better exercise motivation
Patient satisfaction and improvement | Baseline and after 12 weeks of intervention.
  Global Rating of Change Scale will be used for patient satisfaction and to quantify a patient's improvement or deterioration over time to determine the effect of training. Minimally clinically important change is 2 points on 11 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: EBRU CALIK, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No